CLINICAL TRIAL: NCT00000950
Title: Pharmacokinetics of Antituberculosis Agents in HIV-Infected Persons With Tuberculosis
Brief Title: Metabolism of Antituberculosis Drugs in HIV-Infected Persons With Tuberculosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Purpose: Treatment
Other Study IDs: ACTG 309
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2011-03

CONDITIONS: HIV Infections; Tuberculosis
Keywords: Tuberculosis; Isoniazid; Pyrazinamide; Pyridoxine; Rifampin; AIDS-Related Opportunistic Infections; Drug Therapy, Combination; Ethambutol; Acquired Immunodeficiency Syndrome; Antitubercular Agents
MeSH Terms: conditions — HIV Infections; Tuberculosis; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Ethambutol; Isoniazid; Pyrazinamide; Pyridoxine; Rifampin

INTERVENTIONS:
Drug: Ethambutol hydrochloride
Drug: Isoniazid
Drug: Pyrazinamide
Drug: Pyridoxine hydrochloride
Drug: Rifampin

SUMMARY:
The purpose of this study is to determine if a relationship exists between the level of antituberculosis drugs (isoniazid, rifampin, ethambutol, and pyrazinamide) in the blood and the outcome of HIV-positive patients with tuberculosis. This study also evaluates how these drugs are absorbed and metabolized in the body.

DETAILED DESCRIPTION:
Patients receive up to 8 weeks of two or more anti-tuberculosis drugs, of which at least two are isoniazid, rifampin, pyrazinamide, or ethambutol. Blood specimens are collected at 2, 6, and 10 hours after administration of study medication, once between Days 10 and 14 of a phase of daily treatment and once while on an intermittent dose regimen (twice weekly or three times weekly).

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive and have tuberculosis.
* Are 13 years of age or older.
* Have written, informed consent of parent or guardian if you are under 18 years of age.
* Agree to practice abstinence or use barrier methods of birth control during the study.

Exclusion Criteria

You will not be eligible for this study if you:

* Have any other disorder or condition which might cause study treatment to be undesirable.
* Are pregnant.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Primary Completion 2002-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Chirgwin, Study Chair; David Perlman, Study Chair
Locations (13):
- United States (13):
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - Harbor UCLA Med Ctr, Torrance, California
  - University of Miami (Pediatric), Miami, Florida
  - Emory Univ, Atlanta, Georgia
  - Queens Med Ctr, Honolulu, Hawaii
  - Univ of Hawaii, Honolulu, Hawaii
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - SUNY / Health Sciences Ctr at Brooklyn, Brooklyn, New York
  - Beth Israel Med Ctr, New York, New York
  - St Vincent's Hosp / Mem Sloan-Kettering Cancer Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - MetroHealth Med Ctr, Cleveland, Ohio
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Perlman DC, Segal Y, Rosenkranz S, Rainey PM, Peloquin CA, Remmel RP, Chirgwin K, Salomon N, Hafner R; ACTG 309 Team. The clinical pharmacokinetics of pyrazinamide in HIV-infected persons with tuberculosis. Clin Infect Dis. 2004 Feb 15;38(4):556-64. doi: 10.1086/381096. Epub 2004 Jan 28. PMID 14765350